CLINICAL TRIAL: NCT02373345
Title: Clinical and Neuromechanical Predictors for the Evolution of Chronic Non-specific Low Back Pain
Status: Completed | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Institut de Recherche Robert-Sauvé en Santé et en Sécurité du Travail (Other); Chaire de recherche en chiropratique FRCQ (Unknown)
Responsible Party: Principal Investigator, Martin Descarreaux, DC, PhD, Université du Québec à Trois-Rivières
Other Study IDs: UQTR-IRSST-2013-2016
Record Dates: First submitted 2015-02-21; First posted 2015-02-27 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Low Back Pain
Keywords: psychological factors; functional disability; pain thresholds; tolerance thresholds; motor adaptations; natural course
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the present study is to determine the association between factors known to be associated with the development of chronic low back pain (psychological and biological) and the evolution of functional disability in individuals with a history of low back pain. To do so, 100 individuals with a history of nonspecific low back pain will be followed over a period of 18 months. During this time frame, participants will be evaluated three times in the laboratory (initial, at 6 months and at 18 months) to determine pain and tolerance thresholds, pain inhibition processes as well as neuromuscular activation. Moreover, these participants will be assessed every three months (initial, 3, 6, 9 12, 15 and 18 months) for functional disability and pain intensity levels of their low back pain as well as for psychological symptoms usually associated with the development of chronic low back pain. It is hypothesized that high psychological symptoms measured initially will be associated with high functional disability throughout the study .

ELIGIBILITY:
Inclusion Criteria:

* To have experienced at least one episode of disabling (resulting in loss of work or modified tasks at work) nonspecific low back pain in the past three years.

Exclusion Criteria:

* Specific causes of low back pain, arthritic conditions, other chronic pain conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with a history of nonspecific low back pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in disability (Roland-Morris Disability Questionnaire) | baseline, 3 months, 6, months. 9 months, 12 months, 15 months, 18 months
  Roland-Morris Disability Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, DC, PhD, Study Director — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada